CLINICAL TRIAL: NCT05817968
Title: Comparison of a Solid State Versus Balloon Esophageal Catheter for Estimation of Pleural Pressure in Surgical ICU Patients
Brief Title: Solid State vs. Balloon Esophageal Catheter for Estimation of Pleural Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Pulmotech B.V. (Unknown)
Responsible Party: Principal Investigator, Annemijn Jonkman, Assistant Professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MEC-2023-0119
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Failure; Mechanical Ventilation
Keywords: Esophageal manometry; Respiratory monitoring; Mechanical ventilation; Pleural pressure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Method comparison study; participants serve as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal manometry using a solid state sensor vs. balloon catheter (Experimental): Placement of both a solid state and balloon esophageal pressure (Pes) catheter. Pes recordings of these catheters will be acquired simultaneously during both controlled mechanical ventilation and assisted mechanical ventilation, for 10-15 minutes per phase. Ventilator settings/protocol will be as per standard-of-care.
  Interventions: Device: intelligent Esophageal Pressure Catheter (iEPC)

INTERVENTIONS:
Device: intelligent Esophageal Pressure Catheter (iEPC) — Placement of the iEPC nasogastric catheter with solid state sensor for esophageal manometry.
  Comparator: Esophageal balloon catheter (NutriVent).
  Other Names: Solid state esophageal pressure catheter, PulmoTech B.V.

SUMMARY:
Measurements of esophageal pressure (Pes) as surrogate for pleural pressure are routinely performed in selected ICU patients to facilitate lung-protective ventilation and assess breathing effort. Pes is clinically measured via a nasogastric esophageal catheter. Current techniques involve balloon catheters but have some important disadvantages as they could deflate over time and require a very precise positioning and filling volume. A solid-state sensor does not have disadvantages associated with balloon catheters and may therefore be a useful alternative in clinical practice.

This method-comparison study in adult mechanically ventilated ICU patients evaluates the accuracy of Pes measured using an esophageal catheter with a solid-state sensor as compared to a balloon catheter as reference standard.

DETAILED DESCRIPTION:
Measurements of esophageal pressure (Pes) as surrogate for pleural pressure are routinely performed in selected ICU patients to facilitate lung-protective ventilation and assess breathing effort. Pes is clinically measured via a nasogastric esophageal catheter. Current techniques involve balloon catheters but have some important disadvantages as they could deflate over time and require a very precise positioning and filling volume. A solid state sensor does not have disadvantages associated with balloon catheters and may therefore be a useful alternative in clinical practice.

This method-comparison study in adult mechanically ventilated ICU patients evaluates the accuracy of Pes measured using an esophageal catheter with a solid-state sensor as compared to a balloon catheter as reference standard.

Subjects will receive a standard balloon esophageal catheter and a solid-state pressure catheter for simultaneous measurements of Pes. Study population will be post-surgical ICU patients. Measurements will be performed during clinical mechanical ventilation settings which include a first phase of passive controlled ventilation (patient is still sedated after surgery) as well a phase of partially-assisted ventilation where the patient's breathing effort has resumed and is assisted by the ventilator. During both phases, 10-15 minutes of tidal breathing will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient requiring mechanical ventilation at the ICU following cardiothoracic or abdominal surgery
* Age ≥ 18 year

Exclusion Criteria:

* Pregnancy
* Upper airway/esophageal/mouth or face pathology (i.e. recent surgery, esophageal varices, diaphragmatic hernia)
* Nasal bleeding within the last <2 weeks
* Presence of pneumothorax
* Use of anticoagulants that increase the risk of catheter insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Difference in absolute Pes-derived parameters obtained by solid state catheter vs. balloon catheter. | 30 minutes
  Absolute Pes value (in cmH2O) at end-expiration and at peak inspiration (based on flow recordings) will be recorded.
Difference in relative Pes-derived parameters obtained by solid state catheter vs. balloon catheter. | 30 minutes
  Relative Pes value (cmH2O) will be measured as the inspiratory amplitude in Pes.

CONTACTS AND LOCATIONS:
Overall Officials: Annemijn Jonkman, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Oosten JP, Goedendorp N, Mousa A, Flink RC, Schaart R, Flinsenberg M, Somhorst P, Gommers DAMPJ, Heunks L, Jonkman AH. Solid-state esophageal pressure sensor for the estimation of pleural pressure: a bench and first-in-human validation study. Crit Care. 2025 Jan 27;29(1):47. doi: 10.1186/s13054-025-05279-w. PMID 39871347